CLINICAL TRIAL: NCT03305497
Title: Piloting a Naloxone Intervention in an Emergency Response Community to Reduce Opioid Overdoes in Philadelphia
Brief Title: Piloting a Naloxone Intervention in Philadelphia
Status: Completed | Type: Observational
Sponsor: Drexel University (Other)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 1705005398
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Opioids; Harmful Use
Keywords: Opioid Overdose; Naloxone
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Mobile Phone Application — 110 persons will be equipped with a mobile phone application, trained in overdose prevention, and equipped with naloxone. The mobile phone app will allow persons witnessing an overdose to signal persons in the vicinity to respond with naloxone.

SUMMARY:
The escalating opioid overdose epidemic is one of the most serious public health problems confronting the U.S. Death due to drug overdose is a significant and rising cause of mortality and morbidity in Philadelphia. While naloxone is increasingly accessible to combat opioid overdoses, new responses to delivering naloxone to overdose events are needed. The proposed pilot project, to be conducted in Philadelphia, will pursue three specific aims: 1) Identify barriers and facilitators of acceptance and use of a smartphone-based naloxone intervention; 2) Pilot test the implementation of the intervention among 55 non-medical opioid users and 55 community members; 3) Synthesize knowledge acquired in Aims 1 and 2 to be used in a subsequent R01 study to conduct a large-scale, multi-site implementation trial.

DETAILED DESCRIPTION:
The escalating opioid overdose epidemic is one of the most serious public health problems confronting the U.S. In 2014, a record 47,055 people died from a drug overdose in the U.S., which outnumbered deaths from motor vehicle crashes by approximately one and a half times. Heroin and misuse of prescription opioids contributed to a majority of drug overdoses in 2014. Death due to drug overdose is a significant and rising cause of mortality and morbidity in Philadelphia. In 2015, almost 700 drug overdose deaths were reported in Philadelphia - twice as many as deaths from homicide. In response, health policy, legislation, and research funding are increasingly converging in support of the distribution of naloxone, an opioid antagonist, and community-based opioid overdose prevention programs (OPP). The success of OPP is contingent upon the willingness and effectiveness of bystanders to respond to an overdose event and administer naloxone. Emergency Response Communities (ERC) are specialized smartphone-based social networks in which members are approved carriers and/or potential users of a specific medication, such as naloxone. The ERC approach is ideally suited to support, facilitate, and encourage naloxone administration in opioid overdose emergencies, but is untested to date. The model combines GPS and IP-location tracking to identify potential opioid overdose through a smartphone application or app. Towards this end, we are proposing the development and pilot testing of a smartphone app-based naxolone intervention (ERC-NAX) in an ERC in Philadelphia. Research is needed to understand the needs and barriers in communities at high-risk for opioid overdose that will enable effective design, adaption, and implementation of an ERC-NAX app. Guided by preliminary data from study investigators, the proposed pilot project will pursue three specific aims: 1) Identify barriers and facilitators of acceptance and use of a smartphone-based ERC naloxone intervention; 2) Pilot test the implementation of ERC-NAX in an ERC consisting of 55 non-medical opioid users and 55 community members; 3) Synthesize knowledge acquired in Aims 1 and 2 to be used in a subsequent R01 study to conduct a large-scale, multi-site implementation trial. This 3-year study will provide actionable evidence regarding the viability and acceptance of an app-based naloxone intervention following the ERC model. It will be developed and tested in partnership with two community partners in Philadelphia with extensive experience in overdose prevention. This proposed intervention is significant since it leverages the growing success of OPP and will empower communities at high-risk for opioid overdose to provide rapid, secure, and effective emergency response in the event of overdose. This novel intervention, which is designed to augment emergency medical services in the rapid delivery of naloxone to overdose victims, may be effective at deescalating the epidemic of opioid overdose fatalities in Philadelphia and communities elsewhere.

ELIGIBILITY:
Inclusion Criteria:

1. Weekly misuse of heroin and/or rx opioid during past 30 days OR knows active, former, or deceased NMOU 2. Currently lives in zip codes 19122, 19125, 19133, 19134 3. Willingness to carry naloxone 4. Owns smartphone/data package 5. 18 years old or older 6. Speaks/reads English

Exclusion Criteria:

1. Younger than 18
2. Does not speak/read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 55 non-medical users of opioids (NMOU) (e.g., prescription opioids, heroin) and 55 community members who know active, former, or deceased NMOU.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Use of mobile phone app | One year
  Will persons equipped with the mobile phone app signal overdoses and/or respond to overdoses when signaled.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lankenau, PhD, Principal Investigator — Drexel University
Locations (1):
- Kensington, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers.

REFERENCES:
- [Result] Wagner KD, Davidson PJ, Iverson E, Washburn R, Burke E, Kral AH, McNeeley M, Jackson Bloom J, Lankenau SE. "I felt like a superhero": the experience of responding to drug overdose among individuals trained in overdose prevention. Int J Drug Policy. 2014 Jan;25(1):157-65. doi: 10.1016/j.drugpo.2013.07.003. Epub 2013 Aug 9. PMID 23932166
- [Result] Silva K, Schrager SM, Kecojevic A, Lankenau SE. Factors associated with history of non-fatal overdose among young nonmedical users of prescription drugs. Drug Alcohol Depend. 2013 Feb 1;128(1-2):104-10. doi: 10.1016/j.drugalcdep.2012.08.014. Epub 2012 Sep 10. PMID 22974490
- [Result] Lankenau SE, Wagner KD, Silva K, Kecojevic A, Iverson E, McNeely M, Kral AH. Injection drug users trained by overdose prevention programs: responses to witnessed overdoses. J Community Health. 2013 Feb;38(1):133-41. doi: 10.1007/s10900-012-9591-7. PMID 22847602
- [Result] Lankenau SE, Walley A. Opioids and deaths. N Engl J Med. 2011 Feb 17;364(7):686. doi: 10.1056/NEJMc1014490. No abstract available. PMID 21323558
- [Result] Wagner KD, Iverson E, Wong CF, Bloom JJ, McNeeley M, Davidson PJ, McCarty C, Kral AH, Lankenau SE. Personal social network factors associated with overdose prevention training participation. Subst Use Misuse. 2013 Jan;48(1-2):21-30. doi: 10.3109/10826084.2012.720335. Epub 2012 Sep 19. PMID 22988840
- [Derived] Khalemsky M, Khalemsky A, Lankenau S, Ataiants J, Roth A, Marcu G, Schwartz DG. Predictive Dispatch of Volunteer First Responders: Algorithm Development and Validation. JMIR Mhealth Uhealth. 2023 Nov 28;11:e41551. doi: 10.2196/41551. PMID 38015602
- [Derived] Schwartz DG, Ataiants J, Roth A, Marcu G, Yahav I, Cocchiaro B, Khalemsky M, Lankenau S. Layperson reversal of opioid overdose supported by smartphone alert: A prospective observational cohort study. EClinicalMedicine. 2020 Aug 3;25:100474. doi: 10.1016/j.eclinm.2020.100474. eCollection 2020 Aug. PMID 32954238

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT03305497/Prot_SAP_000.pdf